CLINICAL TRIAL: NCT05882747
Title: The Results of Surgery for Renal Cell Carcinoma Metastases in the Pancreas
Brief Title: Renal Cell Carcinoma Metastases to Pancreas
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, carsten palnaes hansen, consultant, DMSC, Rigshospitalet, Denmark
Other Study IDs: RH-2023-3
Record Dates: First submitted 2023-05-21; First posted 2023-05-31 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-05

CONDITIONS: Surgery
Keywords: Pancreatic resection, pancreatic metastase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients' outcome was studied after surgery for renal cell carcinoma. The primary outcome was overall survival and desease free survival. Secondary outcame was complications to surgery.

DETAILED DESCRIPTION:
Study design. The study is a single-center study and includes all patients from the age of 18 who underwent a pancreatic resection due to metastasis from RCC from 1. January 2011 to 31. December 2021. Patients, who underwent additional pancreatic resection after surgery for metastatic RCC, were excluded. The follow-up period ended 31. December 2022.

Data collection. Data are collected from a prospectively maintained database of pancreatic operations, from the electronic hospital record systems Orbit and EPIC, the Danish National Pathology Data Registry, and from the National Register of Death. All Danish Nationals have a unique Central Person Registration number that enables searching of health data.

Outcome. Extracted data included patient demographics, date, and site of nephrectomy, Leibovich score, type of pancreatic resection, 30-days postoperative complications according to the Clavien-Dindo classification system, procedure specific complications (pancreatic fistula or biliary leak) according to the International Study Group on Pancreatic Surgery (ISGPS), pathology of resected pancreatic specimen. Postoperative data included time and site of disease recurrence after pancreatic resection, disease free survival (DS) and overall survival (OS). The postoperative follow-up included standard imaging surveillance with computed tomography scan (CT) of the chest and abdomen at specific intervals depending on the Leibovich score.

Statistics. Clinicopathologic characteristics were summarized using descriptive statistics. Data are presented as median and range if not otherwise stated. Categorial data are presented as numbers or percentage and were analysed with Fisher's exact test. The Kaplan-Meier method was used to estimate survival. Post-pancreatectomy survival was defined as date of pancreatic resection to death. Post-pancreatectomy disease free survival was defined as the median time from the date of pancreatic resection to the date of detection of recurrence of disease, expressed in months. Statistical analysis was performed using GraphPad Version 9.5.1 La Holla, CA. The study was reported according to the STROCSS guidelines.

Ethics The study is a register study and was conducted in accordance with the principles stated in the Declaration of Helsinki. No approval was required according to the Danish National Health Board. The use of register data followed the General Data Protection Regulation of the European Union and was approved by the Danish Data Protection Agency (RH -2015-07, nr. 03616) and patients' consent.

ELIGIBILITY:
Inclusion Criteria: Participants, who underwent pancreatic resection for metastatic renal cell carcinoma -

Exclusion Criteria: Participants, who underwent additional pancreatic resection after surgery for metastatic renal cell carcinoma.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both sex living in Denmark and operated at Rigshospitalet Copenhagen from 1. January 2011 to 31. December 2021.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
overall survival | 1. January 2011 to 31. December 2022
  observational
disease free survival | 1. January 2011 to 31. December 2022
  observational

SECONDARY OUTCOMES:
complications | 1. january 2011 to 31. December 2022
  observational

CONTACTS AND LOCATIONS:
Overall Officials: carsten p hansen, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark

IPD SHARING:
Plan to Share IPD: No
there is no plan to make IPD available

REFERENCES:
- [Background] Saginala K, Barsouk A, Aluru JS, Rawla P, Padala SA, Barsouk A. Epidemiology of Bladder Cancer. Med Sci (Basel). 2020 Mar 13;8(1):15. doi: 10.3390/medsci8010015. PMID 32183076
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204
- [Background] Ballarin R, Spaggiari M, Cautero N, De Ruvo N, Montalti R, Longo C, Pecchi A, Giacobazzi P, De Marco G, D'Amico G, Gerunda GE, Di Benedetto F. Pancreatic metastases from renal cell carcinoma: the state of the art. World J Gastroenterol. 2011 Nov 21;17(43):4747-56. doi: 10.3748/wjg.v17.i43.4747. PMID 22147975
- [Background] Bianchi M, Sun M, Jeldres C, Shariat SF, Trinh QD, Briganti A, Tian Z, Schmitges J, Graefen M, Perrotte P, Menon M, Montorsi F, Karakiewicz PI. Distribution of metastatic sites in renal cell carcinoma: a population-based analysis. Ann Oncol. 2012 Apr;23(4):973-80. doi: 10.1093/annonc/mdr362. Epub 2011 Sep 2. PMID 21890909
- [Background] Sperti C, Pozza G, Brazzale AR, Buratin A, Moletta L, Beltrame V, Valmasoni M. Metastatic tumors to the pancreas: a systematic review and meta-analysis. Minerva Chir. 2016 Oct;71(5):337-44. Epub 2016 Jul 14. PMID 27412234
- [Background] Wiechno P, Kucharz J, Sadowska M, Michalski W, Sikora-Kupis B, Jonska-Gmyrek J, Poniatowska G, Nietupski K, Ossolinski K, Demkow T. Contemporary treatment of metastatic renal cell carcinoma. Med Oncol. 2018 Oct 27;35(12):156. doi: 10.1007/s12032-018-1217-1. PMID 30368624
- [Background] Kalra S, Atkinson BJ, Matrana MR, Matin SF, Wood CG, Karam JA, Tamboli P, Sircar K, Rao P, Corn PG, Tannir NM, Jonasch E. Prognosis of patients with metastatic renal cell carcinoma and pancreatic metastases. BJU Int. 2016 May;117(5):761-5. doi: 10.1111/bju.13185. Epub 2015 Jul 6. PMID 26032863
- [Background] Sun M, Meyer CP, Karam JA, de Velasco G, Chang SL, Pal SK, Trinh QD, Choueiri TK. Predictors, utilization patterns, and overall survival of patients undergoing metastasectomy for metastatic renal cell carcinoma in the era of targeted therapy. Eur J Surg Oncol. 2018 Sep;44(9):1439-1445. doi: 10.1016/j.ejso.2018.05.026. Epub 2018 Jun 5. PMID 29935840
- [Background] Palumbo C, Pecoraro A, Knipper S, Rosiello G, Tian Z, Shariat SF, Simeone C, Briganti A, Saad F, Berruti A, Antonelli A, Karakiewicz PI. Survival and Complication Rates of Metastasectomy in Patients With Metastatic Renal Cell Carcinoma Treated Exclusively With Targeted Therapy: A Combined Population-based Analysis. Anticancer Res. 2019 Aug;39(8):4357-4361. doi: 10.21873/anticanres.13604. PMID 31366530
- [Background] Jaen-Torrejimeno I, Rojas-Holguin A, Lopez-Guerra D, Ramia JM, Blanco-Fernandez G. Pancreatic resection for metastatic renal cell carcinoma. A systematic review. HPB (Oxford). 2020 Apr;22(4):479-486. doi: 10.1016/j.hpb.2019.10.017. Epub 2019 Oct 28. PMID 31672281
- [Background] Anderson B, Williams GA, Sanford DE, Liu J, Dageforde LA, Hammill CW, Fields RC, Hawkins WG, Strasberg SM, Doyle MB, Chapman WC, Khan AS. A 22-year experience with pancreatic resection for metastatic renal cell carcinoma. HPB (Oxford). 2020 Feb;22(2):312-317. doi: 10.1016/j.hpb.2019.05.019. Epub 2019 Jul 23. PMID 31345661
- [Background] Shin TJ, Song C, Jeong CW, Kwak C, Seo S, Kang M, Chung J, Hong SH, Hwang EC, Park JY, Lee H. Metastatic renal cell carcinoma to the pancreas: Clinical features and treatment outcome. J Surg Oncol. 2021 Jan;123(1):204-213. doi: 10.1002/jso.26251. Epub 2020 Oct 12. PMID 33047324
- [Background] Young J, Thompson A, Tait I, Waugh L, McPhillips G. Centralization of services and reduction of adverse events in pancreatic cancer surgery. World J Surg. 2013 Sep;37(9):2229-33. doi: 10.1007/s00268-013-2108-4. PMID 23756771
- [Background] Krautz C, Nimptsch U, Weber GF, Mansky T, Grutzmann R. Effect of Hospital Volume on In-hospital Morbidity and Mortality Following Pancreatic Surgery in Germany. Ann Surg. 2018 Mar;267(3):411-417. doi: 10.1097/SLA.0000000000002248. PMID 28379871
- [Background] Morera-Ocon FJ, Sabater-Orti L, Munoz-Forner E, Perez-Griera J, Ortega-Serrano J. Considerations on pancreatic exocrine function after pancreaticoduodenectomy. World J Gastrointest Oncol. 2014 Sep 15;6(9):325-9. doi: 10.4251/wjgo.v6.i9.325. PMID 25232457
- [Background] Leibovich BC, Blute ML, Cheville JC, Lohse CM, Frank I, Kwon ED, Weaver AL, Parker AS, Zincke H. Prediction of progression after radical nephrectomy for patients with clear cell renal cell carcinoma: a stratification tool for prospective clinical trials. Cancer. 2003 Apr 1;97(7):1663-71. doi: 10.1002/cncr.11234. PMID 12655523
- [Background] Clavien PA, Barkun J, de Oliveira ML, Vauthey JN, Dindo D, Schulick RD, de Santibanes E, Pekolj J, Slankamenac K, Bassi C, Graf R, Vonlanthen R, Padbury R, Cameron JL, Makuuchi M. The Clavien-Dindo classification of surgical complications: five-year experience. Ann Surg. 2009 Aug;250(2):187-96. doi: 10.1097/SLA.0b013e3181b13ca2. PMID 19638912
- [Background] Koch M, Garden OJ, Padbury R, Rahbari NN, Adam R, Capussotti L, Fan ST, Yokoyama Y, Crawford M, Makuuchi M, Christophi C, Banting S, Brooke-Smith M, Usatoff V, Nagino M, Maddern G, Hugh TJ, Vauthey JN, Greig P, Rees M, Nimura Y, Figueras J, DeMatteo RP, Buchler MW, Weitz J. Bile leakage after hepatobiliary and pancreatic surgery: a definition and grading of severity by the International Study Group of Liver Surgery. Surgery. 2011 May;149(5):680-8. doi: 10.1016/j.surg.2010.12.002. Epub 2011 Feb 12. PMID 21316725
- [Background] Bassi C, Marchegiani G, Dervenis C, Sarr M, Abu Hilal M, Adham M, Allen P, Andersson R, Asbun HJ, Besselink MG, Conlon K, Del Chiaro M, Falconi M, Fernandez-Cruz L, Fernandez-Del Castillo C, Fingerhut A, Friess H, Gouma DJ, Hackert T, Izbicki J, Lillemoe KD, Neoptolemos JP, Olah A, Schulick R, Shrikhande SV, Takada T, Takaori K, Traverso W, Vollmer CM, Wolfgang CL, Yeo CJ, Salvia R, Buchler M; International Study Group on Pancreatic Surgery (ISGPS). The 2016 update of the International Study Group (ISGPS) definition and grading of postoperative pancreatic fistula: 11 Years After. Surgery. 2017 Mar;161(3):584-591. doi: 10.1016/j.surg.2016.11.014. Epub 2016 Dec 28. PMID 28040257
- [Background] Blanco-Fernandez G, Fondevila-Campo C, Sanjuanbenito A, Fabregat-Prous J, Secanella-Medayo L, Rotellar-Sastre F, Pardo-Sanchez F, Prieto-Calvo M, Marin-Ortega H, Sanchez-Cabus S, Diez-Valladares L, Alonso-Casado O, Gonzalez-Serrano C, Rodriguez-Sanjuan JC, Garcia-Plaza G, Jaen-Torrejimeno I, Suarez-Munoz MA, Becerra-Massare A, Rio PS, Pando E, Lopez-Andujar R, Munoz-Forner E, Rodriguez-Lopez M, Pereira F, Serrablo-Requejo A, Turrion VS, Garrido MJ, Burdio F, Martin-Perez E, Estevan-Estevan R, Lopez-Guerra D, Castell-Gomez J, Salinas-Gomez J, Lopez-Baena JA, Lopez-Ben S, Solar-Garcia L, Perez-Alonso AJ, Martinez-Insfran LA, Blas JL, Cornejo M, Gutierrez-Calvo A, Pozo CD, Ochando-Cerdan F, Munoz-Bellvis L, Rebollar-Saenz J, Sanchez B, Jover JM, Gomez-Bravo MA, Ramia JM, Rojas-Holguin A. Pancreatic metastases from renal cell carcinoma. Postoperative outcome after surgical treatment in a Spanish multicenter study (PANMEKID). Eur J Surg Oncol. 2022 Jan;48(1):133-141. doi: 10.1016/j.ejso.2021.08.011. Epub 2021 Aug 11. PMID 34417061
- [Background] Malleo G, Salvia R, Maggino L, Marchegiani G, D'Angelica M, DeMatteo R, Kingham P, Pulvirenti A, Sereni E, Jarnagin WR, Bassi C, Allen PJ, Butturini G. Long-term Outcomes After Surgical Resection of Pancreatic Metastases from Renal Clear-Cell Carcinoma. Ann Surg Oncol. 2021 Jun;28(6):3100-3108. doi: 10.1245/s10434-021-09649-w. Epub 2021 Feb 11. PMID 33575870
- [Background] Milanetto AC, Morelli L, Di Franco G, David A, Campra D, De Paolis P, Pasquali C. A Plea for Surgery in Pancreatic Metastases from Renal Cell Carcinoma: Indications and Outcome from a Multicenter Surgical Experience. J Clin Med. 2020 Oct 13;9(10):3278. doi: 10.3390/jcm9103278. PMID 33066168
- [Background] Grassi P, Doucet L, Giglione P, Grunwald V, Melichar B, Galli L, De Giorgi U, Sabbatini R, Ortega C, Santoni M, Bamias A, Verzoni E, Derosa L, Studentova H, Pacifici M, Coppa J, Mazzaferro V, de Braud F, Porta C, Escudier B, Procopio G. Clinical Impact of Pancreatic Metastases from Renal Cell Carcinoma: A Multicenter Retrospective Analysis. PLoS One. 2016 Apr 11;11(4):e0151662. doi: 10.1371/journal.pone.0151662. eCollection 2016. PMID 27064898
- [Background] Benhaim R, Oussoultzoglou E, Saeedi Y, Mouracade P, Bachellier P, Lang H. Pancreatic metastasis from clear cell renal cell carcinoma: outcome of an aggressive approach. Urology. 2015 Jan;85(1):135-40. doi: 10.1016/j.urology.2014.09.034. PMID 25530375
- [Background] Tosoian JJ, Cameron JL, Allaf ME, Hruban RH, Nahime CB, Pawlik TM, Pierorazio PM, Reddy S, Wolfgang CL. Resection of isolated renal cell carcinoma metastases of the pancreas: outcomes from the Johns Hopkins Hospital. J Gastrointest Surg. 2014 Mar;18(3):542-8. doi: 10.1007/s11605-013-2278-2. Epub 2013 Oct 26. PMID 24163138
- [Background] Williamson TJ, Pearson JR, Ischia J, Bolton DM, Lawrentschuk N. Guideline of guidelines: follow-up after nephrectomy for renal cell carcinoma. BJU Int. 2016 Apr;117(4):555-62. doi: 10.1111/bju.13384. Epub 2016 Jan 8. PMID 26617405
- [Background] Ljungberg B, Albiges L, Abu-Ghanem Y, Bedke J, Capitanio U, Dabestani S, Fernandez-Pello S, Giles RH, Hofmann F, Hora M, Klatte T, Kuusk T, Lam TB, Marconi L, Powles T, Tahbaz R, Volpe A, Bex A. European Association of Urology Guidelines on Renal Cell Carcinoma: The 2022 Update. Eur Urol. 2022 Oct;82(4):399-410. doi: 10.1016/j.eururo.2022.03.006. Epub 2022 Mar 26. PMID 35346519
- [Background] Vig SVL, Zan E, Kang SK. Imaging for Metastatic Renal Cell Carcinoma. Urol Clin North Am. 2020 Aug;47(3):281-291. doi: 10.1016/j.ucl.2020.04.005. Epub 2020 Jun 11. PMID 32600531
- [Background] Chiti G, Grazzini G, Cozzi D, Danti G, Matteuzzi B, Granata V, Pradella S, Recchia L, Brunese L, Miele V. Imaging of Pancreatic Neuroendocrine Neoplasms. Int J Environ Res Public Health. 2021 Aug 24;18(17):8895. doi: 10.3390/ijerph18178895. PMID 34501485
- [Background] Raveenthiran S, Esler R, Yaxley J, Kyle S. The use of 68Ga-PET/CT PSMA in the staging of primary and suspected recurrent renal cell carcinoma. Eur J Nucl Med Mol Imaging. 2019 Oct;46(11):2280-2288. doi: 10.1007/s00259-019-04432-2. Epub 2019 Jul 23. PMID 31332498
- [Background] Heidsma CM, Engelsman AF, van Dieren S, Stommel MWJ, de Hingh I, Vriens M, Hol L, Festen S, Mekenkamp L, Hoogwater FJH, Daams F, Klumpen HJ, Besselink MG, van Eijck CH, Nieveen van Dijkum EJ. Watchful waiting for small non-functional pancreatic neuroendocrine tumours: nationwide prospective cohort study (PANDORA). Br J Surg. 2021 Aug 19;108(8):888-891. doi: 10.1093/bjs/znab088. PMID 33783475
- [Background] Sellner F, Thalhammer S, Klimpfinger M. Isolated Pancreatic Metastases of Renal Cell Cancer: Genetics and Epigenetics of an Unusual Tumour Entity. Cancers (Basel). 2022 Mar 17;14(6):1539. doi: 10.3390/cancers14061539. PMID 35326690
- [Background] Azawi NH, Tesfalem H, Mosholt KS, Hoyerup P, Jensen ES, Malchau E, Fode M. Recurrence rates and survival in a Danish cohort with renal cell carcinoma. Dan Med J. 2016 Apr;63(4):A5208. PMID 27034180
- [Background] Piltz S, Meimarakis G, Wichmann MW, Hatz R, Schildberg FW, Fuerst H. Long-term results after pulmonary resection of renal cell carcinoma metastases. Ann Thorac Surg. 2002 Apr;73(4):1082-7. doi: 10.1016/s0003-4975(01)03602-5. PMID 11996245
- [Background] Fottner A, Szalantzy M, Wirthmann L, Stahler M, Baur-Melnyk A, Jansson V, Durr HR. Bone metastases from renal cell carcinoma: patient survival after surgical treatment. BMC Musculoskelet Disord. 2010 Jul 3;11:145. doi: 10.1186/1471-2474-11-145. PMID 20598157
- [Background] Sweeney AD, Fisher WE, Wu MF, Hilsenbeck SG, Brunicardi FC. Retracted: Value of pancreatic resection for cancer metastatic to the pancreas. J Surg Res. 2010 May 15;160(2):268-76. doi: 10.1016/j.jss.2008.04.012. PMID 20422750
- [Background] Santoni M, Conti A, Partelli S, Porta C, Sternberg CN, Procopio G, Bracarda S, Basso U, De Giorgi U, Derosa L, Rizzo M, Ortega C, Massari F, Iacovelli R, Milella M, Di Lorenzo G, Buti S, Cerbone L, Burattini L, Montironi R, Santini D, Falconi M, Cascinu S. Surgical resection does not improve survival in patients with renal metastases to the pancreas in the era of tyrosine kinase inhibitors. Ann Surg Oncol. 2015;22(6):2094-100. doi: 10.1245/s10434-014-4256-7. Epub 2014 Dec 4. PMID 25472645
- [Background] Lyon TD, Roussel E, Sharma V, Carames G, Lohse CM, Costello BA, Boorjian SA, Thompson RH, Joniau S, Albersen M, Leibovich BC. International Multi-institutional Characterization of the Perioperative Morbidity of Metastasectomy for Renal Cell Carcinoma. Eur Urol Oncol. 2023 Feb;6(1):76-83. doi: 10.1016/j.euo.2022.11.003. Epub 2022 Dec 9. PMID 36509653